CLINICAL TRIAL: NCT06359444
Title: Effect of High Intensity Exercise Rehabilitation on Hepatic Fatty Acids (Liver Function), Insulin Sensitivity and Cardiovascular Risk in Patients With MASLD
Brief Title: Effect of High Intensity Exercise Rehabilitation on Liver Function and Insulin Sensitivity in Patients With MASLD
Acronym: CENSORIAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Organization: University Hospital, Ghent (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONZ-2023-0453
Record Dates: First submitted 2024-02-01; First posted 2024-04-11 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Exercise Therapy; Metabolic Dysfunction-associated Steatotic Liver Disease
Keywords: exercise; MASLD; liver diseases
MeSH Terms: conditions — Motor Activity; Liver Diseases | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in two groups: (a) combined aerobic and strength and (b) combined high intensity and strength.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The training will be given by the care provider, but in exercise therapy it is not possible to mask. The assessor will assess the patients without knowing in which group they will be randomized. Randomization will be done by an external person who is only involved for randomization. The investigator, who will be analysing data afterwords, will only see 1 or 2 as group number, but will not know which number is corresponding to which group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined strength + aerobic training (Active Comparator): The patients in this group will exercise for 14 weeks. It is a combination of strength and aerobic exercise.
  Interventions: Other: Combined aerobic + strength training
- Combined strength + HIIT (Experimental): The patients in this group will exercise for 14 weeks. The first 6 weeks consists of combined aerobic and strength exercise, following the protocol from the active comparator group.
  They will switch to combined strength and HIIT exercise for the remaining 8 weeks.
  Interventions: Other: Combined strength + HIIT training

INTERVENTIONS:
Other: Combined aerobic + strength training — Participants will follow a combination of endurance and strength training for 14 weeks.
  There will be three sessions every week: two at Ghent university department of rehabilitation and one at home. Each session will last approximately one hour.
  Arms: Combined strength + aerobic training
Other: Combined strength + HIIT training — 6 weeks of endurance training and strength training, 8 weeks of strength training and HIIT.
  Participants will follow the same combination of endurance and strength training for the first six weeks, to build up to a baseline level of physical fitness. They will then switch to eight weeks of a combination of strength training and High Intensity Interval Training (HIIT).
  There will be three sessions every week: two at Ghent university department of rehabilitation and one at home. Each session will last approximately one hour.
  Arms: Combined strength + HIIT

SUMMARY:
Metabolic dysfunction-associated steatotic liver disease (MASLD) is the most common liver disease worldwide, and is associated with obesity and the metabolic syndrome. Physical activity and lifestyle interventions are among the most recommended treatments for individuals with MASLD.

In this RCT, we will evaluate the effect of combined exercise training "strength and aerobic training" versus "strength and high intensity training (HIIT)". The main outcome parameter is the severity of liver steatosis. Patients will be recruited at the fatty liver clinic of the UZ Gent.

DETAILED DESCRIPTION:
Physical activity and lifestyle interventions, including exercise, are recommended for individuals with metabolic dysfunction-associated steatotic liver disease (MASLD). Weight loss has been found to improve MASLD histologically, but exercise alone can also reduce liver fat accumulation, even without significant weight loss. Exercise has positive effects on chronic inflammation, type 2 diabetes mellitus (T2DM), and mitochondrial function in MASLD patients. Studies suggest that both aerobic and resistance exercise are effective in reducing fat content and liver enzyme levels in MASLD, and thereby generate positive effects on insulin sensitivity and cardiovascular risk. The potential of high-intensity interval training (HIIT) is large in various settings, but was never explored in this population. Moreover, the combination with strength training can have additional health effects which remain to be explored.

All subjects are recruited in the liver steatosis outpatient clinic of the university hospital in Ghent by the physicians and researchers of this study. After patient selection and obtaining informed consent, they will be screened in the rehabilitation center for cardiorespiratory fitness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MASLD by ultrasound, CAP and/or biopsy
* Age between 18 and 75 years old
* No significant liver fibrosis (Fibroscan < 7.5 kPa; if it is between >7.5 and <10, there must be absence of liver fibrosis in the biopsy)

Exclusion Criteria:

* Presence of other liver diseases that may contribute to the clinical presentation in the patient
* Severe cardiovascular, orthopedic, physical or other illnesses that make it impossible to participate in the study's exercise rehabilitation program or where safety cannot be guaranteed
* Pregnancy
* Pharmacological treatment that directly affects MASLD (e.g. GLP-1 analogues)
* A change in medication in the last three months before the study that affects metabolic disease stability

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Liver steatosis by CAP | before training and after training (14 weeks)
  Liver stiffness measurement will be performed using vibration-controlled transient elastography, more specifically the Fibroscan. This method measures the fat accumulation in the liver (dB/m) and the level of scar tissue (kPa), represented as the CAP or steatosis score and the fibrosis score respectively.
Liver steatosis on ultrasound | before training and after training (14 weeks)
  Ultrasound can demonstrate hepatic fatty tissue, estimating severity based on liver-kidney contrast, resolution loss thv the intrahepatic blood vessels, and visibility of the diaphragm. On this basis, a score 0-3 can be assigned.

SECONDARY OUTCOMES:
Insulin sensitivity | before training and after training (14 weeks)
  Insulin sensitivity will be assessed by calculation of the HOMA-IR index (fasting glucose x insulin)
Liver transaminases | before training and after training (14 weeks)
  Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are enzymes located primarily in liver cells. An elevation of these enzymes in the bloodstream may indicate liver damage or inflammation.
Maximal exercise test | before training and after training (14 weeks)
  A ramp protocol will be performed starting at 25 watts, adding 25 watts per minute each time.
  This test will be administered using ergospirometry to derive measures for aerobic physical condition.
Strength | before training and after training (14 weeks)
  Strength will be measured by 1RM determination of the muscle groups that will be trained (leg press, adductors, vertical traction, chest press, abdominal and back muscles). This measurement will be performed at baseline, after 10 weeks and at the end of the study
Cardiovascular function | before training and after training (14 weeks)
  Blood pressure measurements:
  Before and after exercise, systole and diastole blood pressure will be measured. Blood pressure will be measured three times and the average value recorded.
Weight | before training and after training (14 weeks)
  Weight will be measured using a scale to the nearest 0.1 kilogram (kg).
Heigth | before training and after training (14 weeks)
  Height will be measured to the nearest 0.1 meter (m) with a stadiometer.
BMI | before training and after training (14 weeks)
  BMI will be calculated.
waist | before training and after training (14 weeks)
  Waist circumference is measured in standing position with a measuring tape just above the iliac crest, to the nearest 0.1 centimeter (cm).
BIA | before training and after training (14 weeks)
  Bioelectrical impedance analysis (BIA) will be performed to determine lean mass and fat percentage.
Interleukine | before training and after training (14 weeks)
  IL-6 and IL-8 serum levels will be measured in blood. These are correlate with the progression of liver fibrosis and are elevated in patients with chronic liver disease.
TNF-alfa | before training and after training (14 weeks)
  TNF-α is a pro-inflammatory cytokine produced by macrophages and will be measured in blood. Inflammation in NAFLD causes TNF-α to be released into the body. The amount is increased in patients with NAFLD and correlates with the level of fat mass and insulin resistance.
Hepatokines | before training and after training (14 weeks)
  Hepatokines will be measured in blood. These are proteins secreted by the liver which have a demonstrated association with metabolic function/dysfunction. These include fetuin-A, FGF-21, follistatin etc.
Myokines | before training and after training (14 weeks)
  Myokines will be measured in blood. These are proteins secreted by the muscle which have a demonstrated association with metabolic function/dysfunction. These include myostatin, brain-derived neurotrophic factor, etc....
Adipokines | before training and after training (14 weeks)
  Adipokines will be measured in blood. These are proteins secreted by the adipose tissue which have a demonstrated association with metabolic function/dysfunction. These include leptin, adiponectin, etc.
SF-36 | before training and after training (14 weeks)
  Quality of life will be measured using SF-36 (a standard questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Calders, Prof. dr., Principal Investigator — University Ghent; Anja Geerts, Prof. dr., Principal Investigator — University Hospital, Ghent; Sander Lefere, dr., Study Chair — University Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keating SE, Hackett DA, George J, Johnson NA. Exercise and non-alcoholic fatty liver disease: a systematic review and meta-analysis. J Hepatol. 2012 Jul;57(1):157-66. doi: 10.1016/j.jhep.2012.02.023. Epub 2012 Mar 10. PMID 22414768
- [Background] Hashida R, Kawaguchi T, Bekki M, Omoto M, Matsuse H, Nago T, Takano Y, Ueno T, Koga H, George J, Shiba N, Torimura T. Aerobic vs. resistance exercise in non-alcoholic fatty liver disease: A systematic review. J Hepatol. 2017 Jan;66(1):142-152. doi: 10.1016/j.jhep.2016.08.023. Epub 2016 Sep 14. PMID 27639843
- [Background] Oh S, Tsujimoto T, Kim B, Uchida F, Suzuki H, Iizumi S, Isobe T, Sakae T, Tanaka K, Shoda J. Weight-loss-independent benefits of exercise on liver steatosis and stiffness in Japanese men with NAFLD. JHEP Rep. 2021 Feb 10;3(3):100253. doi: 10.1016/j.jhepr.2021.100253. eCollection 2021 Jun. PMID 33898958
- [Background] Karlas T, Petroff D, Sasso M, Fan JG, Mi YQ, de Ledinghen V, Kumar M, Lupsor-Platon M, Han KH, Cardoso AC, Ferraioli G, Chan WK, Wong VW, Myers RP, Chayama K, Friedrich-Rust M, Beaugrand M, Shen F, Hiriart JB, Sarin SK, Badea R, Jung KS, Marcellin P, Filice C, Mahadeva S, Wong GL, Crotty P, Masaki K, Bojunga J, Bedossa P, Keim V, Wiegand J. Individual patient data meta-analysis of controlled attenuation parameter (CAP) technology for assessing steatosis. J Hepatol. 2017 May;66(5):1022-1030. doi: 10.1016/j.jhep.2016.12.022. Epub 2016 Dec 28. PMID 28039099

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/44/NCT06359444/SAP_000.pdf